CLINICAL TRIAL: NCT05473806
Title: Prospective, Multicenter, Randomized, and Comparative Clinical Trials to Compare the Effects of Pioglitazone and Evogliptin on Hepatic Fibrosis in Patients With Chronic Hepatitis B With Significant Hepatic Fibrosis With Type 2 Diabetes
Brief Title: Effects of Pioglitazone and Evogliptin on Hepatic Fibrosis in Patients With Chronic Hepatitis B With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seung Up Kim (Other)
Responsible Party: Sponsor-Investigator, Seung Up Kim, professor, Yonsei University
Organization: Yonsei University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-DASU-01
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B, Chronic; Fibrosis, Liver; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis; Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Tablets; 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pioglitazone 15mg (Experimental): pioglitazone hydrochloride. PO. 2 tablets once a day.
  Interventions: Drug: Pioglitazone 15 Mg Oral Tablet
- Evogliptin 5mg (Experimental): Evogliptin tartrate. PO. 1 tablets once a day.
  Interventions: Drug: Evogliptin 5mg

INTERVENTIONS:
Drug: Pioglitazone 15 Mg Oral Tablet — 24weeks dose
  Other Names: Gluconon tablet 15mg
  Arms: Pioglitazone 15mg
Drug: Evogliptin 5mg — 24weeks dose
  Other Names: SUGANON tablet 5mg
  Arms: Evogliptin 5mg

SUMMARY:
An exploratory comparison of changes in liver fibrosis through glycemic control within and between groups after administration of Pioglitazone and Evogliptin in chronic hepatitis B patients with type 2 diabetes and liver fibrosis

DETAILED DESCRIPTION:
Subjects who satisfy the selection/exclusion criteria and agree to participate in the clinical trial are randomly assigned to receive clinical trial drugs in a 1:1 ratio based on Visit 2 (Baseline) and take it for 24 weeks.

After that, visits are made at 12 and 24 weeks, and necessary tests are performed to confirm the improvement of liver fibrosis and to evaluate safety.

[Number of subjects and basis for calculation] The target number of test subjects is 40 in total, with 20 in each group (including 10% dropout rate).

The study design is an interventional study design comparing two test drugs, and it is intended to be performed as an exploratory study on safety and efficacy to confirm the possibility of entering a therapeutic confirmation trial.

The number of subjects was assumed by referring to the study on the measurement of liver fibrosis in NAFLD patients with type 2 diabetes in Reference which was conducted as hepatitis B patients with type 2 diabetes, the target disease of this clinical trial.

Significance level: 0.05 (two-sided test) statistical power: 90% Difference in the amount of change before and after treatment: 3.7 Standard deviation: 4.416324172 (Utilizing previous research results, the standard deviation of the difference was calculated by calculating the inverse function of the t distribution.)

G-power was used to calculate the number of subjects, and since this study is an exploratory comparative study between two groups and two independent groups, 18 people are needed per group, so a total of 36 people are needed. Considering dropout of about 10%, a total of 40 subjects, 20 in each group, will participate in this study.

[randomization] Randomization is based on a randomization table previously generated by a medical statistician. Therefore, the suitability of the subject is judged before the subject is randomly assigned to the two groups. Randomization will be conducted at a ratio of 1:1 to Test Group 1 and Test Group 2, respectively, based on the number of subjects for each clinical trial participating institution.

During clinical trial registration, subjects who have signed the consent form can only be identified with a unique subject identification code given to each subject instead of their name, and a random number will be continuously assigned by the researcher.

The randomization number is determined according to a computer-generated randomization code, and the randomization number determines the study drug group for the subject.

Randomization numbers are assigned sequentially according to the order of subject registration, and subjects will be continuously supplied with drugs based on the same dosing number during the clinical trial period.

Each Principal Investigator or Investigator shall check the randomization number assigned to each subject whenever a subject is enrolled in serial number order, and then start administration of the study drug accordingly. If a subject withdraws from the clinical trial, the randomization number assigned to the subject cannot be reused, and the subject cannot participate again in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 20 or over and under 80 years of age
* Those who satisfy the following conditions among chronic hepatitis B patients diagnosed with type 2 diabetes.

first. For the first diagnosis of type 2 diabetes: 6.5% ≤ HbA1c < 10.0%; second. Diagnosed with type 2 diabetes: HbA1c < 10.0%;

* Subjects who show significant liver fibrosis of 7 kilopascal or more in liver elasticity test using Fibroscan.
* Subjects who voluntarily sign the informed consent form after understanding the clinical study and being informed of the risks and benefits.

Exclusion Criteria:

* Those who are currently taking Pioglitazone or Evogliptin, or those who have stopped taking medication for less than 4 weeks.
* Patients meeting the criteria for alcoholic fatty liver (if alcohol intake exceeds 210 g per week for men and 140 g per week for women for the past 2 years)
* Cirrhosis patients with decreased liver function (CTP class B and C)
* Those taking drugs that can cause fatty liver (amiodarone, methotrexate, tamoxifen, valproate, corticosteroids, etc.)
* Patients with acute or chronic metabolic acidosis, including diabetic ketoacidosis with or without coma, and patients with a history of ketoacidosis (within 24 weeks)
* In case of allergy or hypersensitivity reaction to the target drug or its components.
* Patients treated with oral or parenteral corticosteroids chronically (>14 consecutive days) within 8 weeks prior to screening
* Malnutrition, starvation, and debilitating conditions (including patients with severe infections and severe trauma before and after surgery)
* Patients receiving or receiving radiation and chemotherapy for malignancy for less than 2 years.
* Heart failure (class III-IV in New York Heart Association classification) or uncontrolled arrhythmias within 24 weeks

table. New York Heart Association Classification. Class I: Normal athletic ability; Class Ⅱ: Difficulty breathing, palpitations, chest pain, etc. appear due to daily exercise (fast walking or climbing a hill); Class Ⅲ: Symptoms appear with light exercise (walking on flat ground); Class IV: Symptoms appear even at rest;

* Patients with acute cardiovascular disease within 12 weeks (patients with a history of unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass graft, or coronary intervention)
* Patients with renal failure, chronic renal disease (estimated glomerular filtration rate <60 mL/min/1.73 m2) or patients on dialysis.
* Anemic patients with an Hb level of less than 10.5 g/dl.
* Pregnant or lactating women
* Patients who do not consent to the use of appropriate contraceptive methods during the clinical trial period only for women or men of childbearing potential.
* Patients who have taken clinical trial drugs from other clinical trials within 4 weeks of consenting to the document.
* Persons unable to participate in clinical trials due to the judgment of other researchers.
* Persons who cannot read consent forms (eg illiterate, foreigners, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2023-02-19 (Estimated)

PRIMARY OUTCOMES:
Changes in Liver Stiffness Measurement at 24 weeks compared to baseline. | 24 weeks
  It is measured based on the CAP score(db/m) and kilopascal from the liver fibroscan and evaluated by performing the paired-sample t-test or Wilcoxon signed test.

SECONDARY OUTCOMES:
Changes in Controlled Attenuation Parameter(CAP) value at 24 weeks compared to baseline. | 24 weeks
  The rate of decrease in the amount of fatty liver (CAP Value) measured at the end of the evaluation compared to the baseline is a descriptive statistic defined as [(Baseline CAP Value)- (Follow-up CAP Value)] / (Baseline CAP Value) × 100 (%) (mean, standard deviation, median, range (minimum, maximum)) are presented.
Changes in HbA1c at 24 weeks compared to baseline. | 24 weeks
  After 24 weeks of treatment, the degree of change in HbA1c compared to baseline is defined as absolute difference = [= (Baseline HbA1c)-(Follow-up HbA1c)] and evaluated by performing paired-sample t-test or Wilcoxon signed-rank test.
Changes in Insulin at 24 weeks compared to baseline. | 24 weeks
  After 24 weeks of treatment, the degree of change in Insulin compared to baseline is defined as absolute difference = [= (Baseline Insulin)-(Follow-up Insulin)] and evaluated by performing paired-sample t-test or Wilcoxon signed-rank test.
Changes in lipid profile at 24 weeks compared to baseline. | 24 weeks
  After 24 weeks of treatment, the degree of change in lipid profile compared to baseline is defined as absolute difference = [= (Baseline lipid profile)-(Follow-up lipid profile)] and evaluated by performing paired-sample t-test or Wilcoxon signed-rank test.
Changes in aspartate aminotransferase(AST)/alanine aminotransferase(ALT) at 24 weeks compared to baseline. | 24 weeks
  It is evaluated by performing paired-sample t-test or Wilcoxon signed rank test.
  The proportion of subjects whose aspartate aminotransferase(AST)/alanine aminotransferase(ALT) recovered to normal values compared to baseline was Frequency and percentages are given and assessed using either the chi-square test or Fisher's exact test.
Changes in Body weight at 24 weeks compared to baseline. | 24 weeks
  It is evaluated by performing paired-sample t-test or Wilcoxon signed rank test.
Rate of side effects and discontinuation or change of drug after 24 weeks compared to baseline | 24 weeks
  It is evaluated by performing paired-sample t-test or Wilcoxon signed rank test.
Analysis of predictors of improvement in liver fibrosis after 24 weeks compared to baseline. | 24 weeks
  It is analyzed the subject's fibroscan(CAP score(db/m) and kilopascal), body weight, aminotransferase(AST)/alanine aminotransferase(ALT), lipid profile, hepatitis serum markers(Hepatitis B surface antigen(HBsAg),Hepatitis B e-antigen(HBeAg),Anti-Hepatitis B e-antigen(Anti-HBe),Anti-Hepatitis B surface antigen(Anti-Hbs),Anti-hepatitis C virus(Anti-HCV)), drug compliance.
Analysis of predictors of improvement of fatty liver after 24 weeks compared to baseline. | 24 weeks
  It is analyzed the subject's fibroscan(CAP score(db/m) and kilopascal), body weight, aminotransferase(AST)/alanine aminotransferase(ALT), lipid profile, hepatitis serum markers(Hepatitis B surface antigen(HBsAg),Hepatitis B e-antigen(HBeAg),Anti-Hepatitis B e-antigen(Anti-HBe),Anti-Hepatitis B surface antigen(Anti-Hbs),Anti-hepatitis C virus(Anti-HCV)), drug compliance.
Analysis of predictors of HbA1c improvement after 24 weeks compared to baseline. | 24 weeks
  It is analyzed the subject's fibroscan(CAP score(db/m) and kilopascal), body weight, Homeostatic Model Assessment for Insulin Resistance, drug compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Up Kim, Principal Investigator — Severance Hospital
Locations (4):
- South Korea (4):
  - Gangnam Severance Hospital, Seoul
  - Samsung seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul